CLINICAL TRIAL: NCT05566249
Title: A Study to Validate the Safety and Feasibility of ArtiSential in Colorectal Cancer Surgery Using Prospectively Constructed Multi-center Registry
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Seoul St. Mary's Hospital (Other); Chonnam National University Hospital (Other); Severance Hospital (Other); Seoul National University Bundang Hospital (Other); Uijeongbu St. Mary Hospital (Other); LivsMed (Unknown)
Responsible Party: Principal Investigator, Jung Wook Huh, Professor, Samsung Medical Center
Other Study IDs: SMC-2022-01-174
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer; Rectosigmoid Cancer; Rectosigmoid Junction Cancer
Keywords: laparoscopic surgery; minimally invasive surgery; robotic-assisted surgery; robotic surgery; Da Vinci system; ArtiSential; Articulating laparoscopic instrument
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ArtiSential group: Patients undergoing laparoscopic surgery using ArtiSential
  Interventions: Device: ArtiSential
- Robot group: Patients undergoing robotic surgery

INTERVENTIONS:
Device: ArtiSential — Articulating laparoscopic instrument
  Groups: ArtiSential group

SUMMARY:
This study is to validate the safety and feasibility of ArtiSential (Articulating laparoscopic instrument) colorectal surgery and compare it with robotic surgery for patients with rectal cancer and rectosigmoid junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 ~ 80 year old male or female
* Biopsy-proven adenocarcinoma
* Rectal cancer or Rectosigmoid junction cancer
* Primary cancer
* Non-metastatic cancer
* Planned (or elective) curative resection
* Low anterior resection with double-stapled technique

Exclusion Criteria:

* Preoperative systemic chemotherapy
* Distant metastasis at initial diagnosis
* Palliative surgery
* Emergent surgery
* Lynch syndrome or FAP-associated cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with rectal or rectosigmoid junction adenocarcinoma who will be planned to undergo elective low anterior resection with double stapled technique.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical failure | 1 month
  conversion, postoperative complications, or less than 12 harvested lymph nodes
Cost | 1 month
  Total medical cost during hospital stay for surgery

SECONDARY OUTCOMES:
Oncologic outcomes | 5-year
  5-year Disease-free Survival
Oncologic outcomes | 5-year
  5-year Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Pyo DH, Kim S, Do M, Huh JW. Laparoscopic Ultralow Anterior Resection Using a New Articulating Device. Dis Colon Rectum. 2025 Jan 1;68(1):e5. doi: 10.1097/DCR.0000000000003287. Epub 2024 Sep 12. No abstract available. PMID 39264062